CLINICAL TRIAL: NCT06170359
Title: The Effect of Preemptive Administration of Pregabalin on Postoperative Pain and Respiratory Dynamics in Patients Undergoing Surgery for Robotic Radical Prostatectomy.
Brief Title: The Effect of Preemptive Pregabalin on Postoperative Pain and Respiratory Dynamics in Robotic Prostatectomy Operation.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Senay Goksu, SPECIALIST, MD,, Umraniye Education and Research Hospital
Other Study IDs: Preemptive Pregabalin
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Pain, Acute
Keywords: preemptive analgesia, pregabalin, pain, robotic surgery
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: those who did not take pregabalin (n:45)
  Interventions: Procedure: robotic surgery under general anaesthesia
- Group 2: those who took pregabalin (n:45)
  Interventions: Procedure: robotic surgery under general anaesthesia

INTERVENTIONS:
Procedure: robotic surgery under general anaesthesia — During robotic surgery, the standard 45-degree upright Trendelenburg position and for postoperative analgesia, 0.06 mg/kg morphine, 1 gram (g) paracetomol and 8 mg onasetron are administered iv to all patients 30 minutes before the end of the operation. At the end of surgery and after extubation, patients are taken from the recovery unit to the service. In the service, all patients are given paracetamol 1g every 8 hours and tenoxicam 20 mg every 24 hours for pain treatment. Tramadol 1 mg/kg iv is administered as rescue analgesic to patients with a VAS score >4.

SUMMARY:
The study aimed to investigate the impact of preemptive pregabalin on the postoperative pain severity and the requirement of analgesic drugs in patients undergoing robotic radical prostatectomy surgery as primary outcome.

Additionally, it examined the effect of pregabalin on early postoperative respiratory dynamics as secondary outcome.

DETAILED DESCRIPTION:
Our study will be conducted on a total of 90 patients after ethics committee approval and patient consent. In the prospective observational study, patients will be divided into two groups: those who received preoperative pregabalin and those who did not.

Group 1: those who did not take pregabalin (n:45) Group 2: those who took pregabalin (n:45) Procedure to be applied (interventions) Those who have received pregabalin treatment drink 150 mg of pregabalin with a small amount of water 2 hours before the surgical procedure. All patients receive standard general anesthesia in the operating room after standard hemodynamic monitoring, invasive arterial pressure and Bispectral Index (BIS) monitoring.

Afterwards, all patients receive standard anesthesia maintenance and are monitored in mechanical ventilation (volume-controlled mode), PEEP at 7-8 cmH20 and ETCO2 level at 30-35mmHg during the pneumoperitoneum period. During the pneumoperitoneum period, intra-abdominal pressure is kept within the range of 12-14 mmHg.

During robotic surgery, the standard 45-degree upright Trendelenburg position and perioperative restrictive fluid management are performed. For postoperative analgesia, 0.06 mg/kg morphine, 1 gram (g) paracetomol and 8 mg onasetron are administered iv to all patients 30 minutes before the end of the operation. At the end of surgery and after extubation, patients are taken from the recovery unit to the service in accordance with Aldrete criteria. In the service, all patients are given paracetamol 1g every 8 hours and tenoxicam 20 mg every 24 hours for pain treatment. Tramadol 1 mg/kg iv is administered as rescue analgesic to patients with a VAS score >4.

Recording Data Patients' age, gender, BMI, and comorbidities are recorded. Perioperative heart rate (HR), mean arterial pressure (MAP), peripheral oxygen saturation (SpO2), BIS value, ETCO2, PaCO2 (arterial blood gas), PaO2/Fi02 and peak airway pressure (Ppeak), plateau pressure (Pplato). ) is recorded at the times specified below.

T0: 10th minute after anesthesia induction (supine position 00) T1: 10 minutes after the start of pneumoperitoneum (supine position 00) T2: 30 minutes after the upright Trendelenburg position (450) T3: At the end of pneumoperitoneum (supine position 00) T4: 30 minutes after extubation (recovery unit) The FEV1, FVC, FEV1/FVC values of all patients in the routine respiratory function test performed preoperatively and on the second postoperative day are recorded.

Operation time, Trendelenburg time, perioperative urine amount and general fluid balance are recorded.

Postoperative pain levels of all patients were 30 minutes and 6, 12, 24, 36 days after extubation. It is evaluated and recorded with VAS (Visual Analog Scale) between 0-10 at the 48th and 48th hours.

Analgesic medications administered postoperatively, time of first rescue analgesic (tramadol) administration, total tramadol consumption amount, presence of nausea-vomiting, dizziness, visual impairment, presence of upper airway problems, pulmonary and surgical complications are recorded.

ELIGIBILITY:
Inclusion Criteria:

Patients between the ages of 18-75 and with an ASA score of 1-3 who will undergo robotic radical prostatectomy (RARP) surgery under general anesthesia Exclusion criteria Under 18 years of age, over 75 years of age, ASA over 3, history of severe COPD and asthma, history of lobectomy/pneumonectomy, restrictive lung disease, congestive heart failure (NYHA stage 3-4), severe renal and hepatic dysfunction, history of neuromuscular disease, neurological and those with psychiatric problems, extreme obesity or malnutrition (Body mass index >30 or <20), chronic alcohol and opioid use, gabapentinoid, opioid allergy or intolerance, history of chronic pain or fibromyalgia, history of malignant neoplasm, history of gastrointestinal bleeding or perforation, patients in need of intensive care and those who do not consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-75 and with an ASA score of 1-3 who will undergo robotic radical prostatectomy (RARP) surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
To investigate the impact of preemptive pregabalin on the postoperative pain | 5 times during surgery and up to 48 hours after surgery
  to investigate the impact of preemptive pregabalin on the postoperative pain severity and the requirement of analgesic drugs in patients undergoing robotic radical prostatectomy surgery

SECONDARY OUTCOMES:
the effect of pregabalin on early postoperative respiratory dynamics | 5 times during surgery and up to 48 hours after surgery
  we will examine the effect of pregabalin on early postoperative respiratory dynamics

IPD SHARING:
Plan to Share IPD: No